CLINICAL TRIAL: NCT01638546
Title: A Multi-Center, Randomized, Double-Blind Phase II Study Comparing ABT-888, a PARP Inhibitor, Versus Placebo With Temozolomide in Patients With Relapsed Sensitive or Refractory Small Cell Lung Cancer
Brief Title: Temozolomide With or Without Veliparib in Treating Patients With Relapsed or Refractory Small Cell Lung Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NCI-2012-01130; NCI-2012-01130 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000737062; 12-021; IRB #12-021; 9026 (Other: Memorial Sloan Kettering Cancer Center); 9026 (Other: CTEP); N01CM00039 (NIH); P30CA008748 (NIH); U01CA070095 (NIH); UM1CA186691 (NIH)
Record Dates: First submitted 2012-07-09; First posted 2012-07-11 (Estimated); Results first posted 2018-03-27 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-09

CONDITIONS: Recurrent Lung Small Cell Carcinoma
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Temozolomide; veliparib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (veliparib and temozolomide) (Experimental): Patients receive veliparib PO BID on days 1-7 and temozolomide PO on days 1-5.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Temozolomide; Drug: Veliparib
- Arm II (placebo and temozolomide) (Active Comparator): Patients receive placebo PO BID on days 1-7 and temozolomide as in Arm I.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Placebo Administration; Drug: Temozolomide

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Placebo Administration — Given PO
  Arms: Arm II (placebo and temozolomide)
Drug: Temozolomide — Given PO
  Other Names: CCRG-81045; Gliotem; Imidazo[5,1-d]-1,2,3,5-tetrazine-8-carboxamide, 3, 4-dihydro-3-methyl-4-oxo-; M & B 39831; M and B 39831; Methazolastone; RP-46161; SCH 52365; Temcad; Temizole; Temodal; Temodar; Temomedac; TMZ
Drug: Veliparib — Given PO
  Other Names: ABT 888; ABT-888; ABT888; PARP-1 inhibitor ABT-888
  Arms: Arm I (veliparib and temozolomide)

SUMMARY:
This randomized phase II trial studies how well temozolomide with or without veliparib works in treating patients with small cell lung cancer that has returned or does not respond to treatment. Temozolomide works by damaging molecules inside the cancer cells, such as deoxyribonucleic acid (DNA), that are needed for cancer survival and growth. Veliparib may stop the growth of tumor cells by blocking proteins that are needed for repairing the damaged DNA and it may also help temozolomide to kill more cancer cells. It is not yet know whether temozolomide is more effective with or without veliparib in treating patients with relapsed or refractory small cell lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To demonstrate an improvement in progression free survival (PFS) at four months in patients with relapsed sensitive or refractory small cell lung cancer (SCLC) receiving ABT-888 (veliparib) and temozolomide compared to placebo and temozolomide.

SECONDARY OBJECTIVES:

I. Determine the objective response rate (ORR) (based on Response Evaluation Criteria in Solid Tumors [RECIST] 1.1 criteria) in both arms of the study: ABT-888 and temozolomide and placebo and temozolomide.

II. Determine the overall survival (OS) of patients in both arms of the study. III. Determine the ORR, PFS and OS of ABT-888 and temozolomide and placebo and temozolomide, in the following patient groups: sensitive disease vs. refractory disease; second-line treatment vs. third-line treatment; brain metastases vs. no brain metastases.

IV. Determine the safety and tolerability of ABT-888 and temozolomide in patients with SCLC.

TERTIARY OBJECTIVES:

I. Evaluate available tumor samples for methylated O6-methylguanine-DNA methyltransferase (MGMT) promoter by the EpiTyper assay, as well as MGMT expression by immunohistochemistry and determine if these correlate with PFS, ORR, and OS.

II. Evaluate available tumor samples for poly (ADP ribose) polymerase (PARP)-1, breast cancer 1 (BRCA-1) and RAD51 recombinase (RAD51) expression by immunohistochemistry and determine if they correlate with PFS, ORR, and OS.

III. Evaluate available tumor samples for messenger ribonucleic acid (mRNA) BRCA-1 expression and determine if it correlates PFS, ORR, and OS.

IV. Evaluate available tumor samples for phosphatase and tensin homolog (PTEN) expression by immunohistochemistry and determine if it correlates PFS, ORR, and OS.

V. Identify and enumerate circulating tumor cells (CTCs) using the Cell Search System in these patients with SCLC at baseline and at the time of repeat imaging.

VI. Correlate the number of CTCs with PFS and OS at each time point. VII. Correlate the change in CTCs with radiographic response. VIII. Correlate the number of CTCs at baseline with patient characteristics (disease burden, location of metastases, progression at existing sites or new sites of disease).

IX. Evaluate gamma H2A histone family, member X (H2AX)-positive CTCs using the CellSearch.

X. Assess the percentage increase in DNA fragments during treatment and correlate with outcome in each of the treatment groups.

XI. Evaluate plasma markers for apoptosis and angiogenesis. XII. Assess changes in plasma markers for apoptosis and angiogenesis, including caspase-cleaved cytokeratin 18 fragment (M30), soluble cytokeratin 18 (M65), pro-gastrin-releasing peptide (pro-GRP), soluble vascular endothelial growth factor (sVEGF), sVEGF receptor 2 (sVEGFR2), and soluble v-kit Hardy-Zuckerman 4 feline sarcoma viral oncogene homolog (sKIT), and correlate these markers with outcome in the two treatment arms.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive veliparib orally (PO) twice daily (BID) on days 1-7 and temozolomide PO on days 1-5.

ARM II: Patients receive placebo PO BID on days 1-7 and temozolomide as in Arm I.

In both arms, courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 8-12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed small cell lung cancer; confirmation will be done at Memorial Sloan-Kettering Cancer Center (MSKCC) or locally for participating sites
* Patients' disease has relapsed or progressed after one or two prior chemotherapy regimens, one of which must have been an etoposide-platinum doublet; eligible patients will be defined as follows:

  * "Sensitive" disease: patients who had one previous line of chemotherapy and maintained an appropriate response for > 60 days
  * "Refractory" disease: those patients with either (a) no response to first-line chemotherapy or progression =< 60 days after completing treatment, or (b) "sensitive" or "refractory" disease in need of third-line therapy (i.e. completed or failed two previous lines of chemotherapy)
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1 (Karnofsky >= 70%)
* Patients with asymptomatic brain metastases that do not require immediate whole brain radiation therapy and are on stable doses of steroids are allowed
* Patients must have measurable disease, which is defined as at least one lesion that can be accurately measured in at least one dimension on a computed tomography (CT) scan as per RECIST version 1.1; brain metastases can be considered measurable disease if they meet this criterion
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Hemoglobin >= 8.5 g/dL; the use of transfusion to achieve this criterion should be at the discretion of the investigators
* Total bilirubin =< 1.5 mg/dL x institutional upper limit of normal
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3.0 x institutional upper limit of normal
* Creatinine =< 1.5 x institutional upper limit of normal OR creatinine clearance >= 50 mL/min/1.73 m^2 for patients with creatinine levels >= 1.5 x upper limit of institutional normal
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* For women of child-bearing potential, negative pregnancy test within 14 days prior to starting temozolomide and ABT-888
* Ability to understand and the willingness to sign a written informed consent document
* Able to swallow pills
* Patients will not be excluded based on the diagnosis of acquired immune deficiency syndrome (AIDS); given the increased risk of infection, these patients should have cluster of differentiation (CD)4 counts above 200 cells/mm^3; patients with AIDS or human immunodeficiency virus (HIV) not receiving agents with the potential for pharmacokinetic interactions with ABT-888 may be eligible

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 3 weeks prior to entering the study
* Patients who have not recovered from adverse events due to agents administered more than 3 weeks earlier; toxicities should have resolved to baseline or to within one grade level of their baseline (not to exceed grade 2)
* Patients who have been administered ABT-888, any other PARP-inhibitor, or temozolomide
* Patients may not be receiving any other investigational agents
* Patients with leptomeningeal involvement
* Patients with active seizures or a history of seizures
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to ABT-888 or temozolomide
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with ABT-888; these potential risks also apply to temozolomide
* Patients with either AIDS or HIV on combination antiretroviral therapy are ineligible
* Patients with a synchronous active malignancy requiring treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2012-07-27 (Actual); Primary Completion 2017-01-09 (Actual); Study Completion 2026-03-25 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Charles M Rudin, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (14):
- United States (14):
  - Moffitt Cancer Center, Tampa, Florida
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Washington University School of Medicine, St Louis, Missouri
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Sleepy Hollow, Sleepy Hollow, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Case Western Reserve University, Cleveland, Ohio
  - M D Anderson Cancer Center, Houston, Texas
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia

REFERENCES:
- [Derived] Pietanza MC, Waqar SN, Krug LM, Dowlati A, Hann CL, Chiappori A, Owonikoko TK, Woo KM, Cardnell RJ, Fujimoto J, Long L, Diao L, Wang J, Bensman Y, Hurtado B, de Groot P, Sulman EP, Wistuba II, Chen A, Fleisher M, Heymach JV, Kris MG, Rudin CM, Byers LA. Randomized, Double-Blind, Phase II Study of Temozolomide in Combination With Either Veliparib or Placebo in Patients With Relapsed-Sensitive or Refractory Small-Cell Lung Cancer. J Clin Oncol. 2018 Aug 10;36(23):2386-2394. doi: 10.1200/JCO.2018.77.7672. Epub 2018 Jun 15. PMID 29906251

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm II (Placebo and Temozolomide): Patients receive placebo PO BID on days 1-7 and temozolomide as in Arm I.
  Laboratory Biomarker Analysis: Correlative studies
  Placebo: Given PO
  Temozolomide: Given PO
Period: Overall Study
Arm/Group | Arm I (Veliparib and Temozolomide) | Arm II (Placebo and Temozolomide)
Started | 52 | 45
Completed | 51 | 42
Not Completed | 1 | 3
Not completed — Adverse Event | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Veliparib and Temozolomide) | Arm II (Placebo and Temozolomide) | Total
Number analyzed (Participants) | 52 | 45 | 97
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 31 | 31 | 62
  >=65 years | 21 | 14 | 35
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 23 | 52
  Male | 23 | 22 | 45
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 1 | 5
  White | 47 | 43 | 90
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival, Calculated as the Proportion of Patients Alive and Without Evidence of Disease
Description: Compared across the two arms using a Fisher exact test.
Time Frame: From randomization to time of progression or death, whichever occurs first, assessed at 4 months
Measure: Number; unit: participants
Arm/Group | Arm I (Veliparib and Temozolomide) | Arm II (Placebo and Temozolomide)
Number analyzed (Participants) | 51 | 42
participants | 18 | 11
Statistical Analysis 1: Comparison: Arm I (Veliparib and Temozolomide) vs Arm II (Placebo and Temozolomide); Test type: Other; The study will be performed as a double-blind, placebo controlled, randomized Phase II in patients with relapsed sensitive or refractory SCLC. Eligible patients will be randomized 1:1 to one of two treatment arms: ABT-888 and temozolomide as the investigational arm, versus placebo and temozolomide as the control arm. The randomization will be stratified by center and by type or relapse (sensitive vs. refractory). The primary objective is to compare the two treatment regimens with respect to efficacy, expressed as Progression Free Survival (PFS) at 4 months post-randomization. PFS will be calculated as proportion of patients alive and without evidence of disease at 4 months after randomization

2. Secondary Outcome: Overall Response (ORR) by RECIST 1.1 Criteria
Description: Corresponding exact two-sided 95% confidence intervals will be calculated and reported in both arms of the study. Comparisons between treatment arms will be performed using Fisher-exact test.
Time Frame: From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 4 months
Measure: Number; unit: participants
Arm/Group | Arm I (Veliparib and Temozolomide) | Arm II (Placebo and Temozolomide)
Number analyzed (Participants) | 51 | 42
participants | 20 | 6

3. Secondary Outcome: Overall Survival
Description: Estimated in each treatment group using Kaplan-Meier method. Group comparisons will be performed using log-rank test.
Time Frame: From randomization to time of death
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (Veliparib and Temozolomide) | Arm II (Placebo and Temozolomide)
Number analyzed (Participants) | 51 | 42
months | 8.2 [6.4 to 12.2] | 7 [5.3 to 9.5]

4. Secondary Outcome: Number of Participants With Adverse Events
Description: Tabulated According to the National Cancer Institute Common Terminology Criteria for Adverse Events Version 4.0. Summary level.
Time Frame: From the start of treatment until 30 days from coming off treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Veliparib and Temozolomide) | Arm II (Placebo and Temozolomide)
Number analyzed (Participants) | 52 | 45
Participants | 52 | 45

5. Other Pre Specified Outcome: BRCA1 Expression, Assessed by Immunohistochemistry
Description: Fisher's exact test will be used to correlate response and log-rank test to correlate with progression free survival and overall survival.
Time Frame: Up to 5 years
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Changes in Plasma Markers
Description: Correlated with outcome in the two treatment arms.
Time Frame: Baseline to up to 5 years
Reporting Status: Not Posted

7. Other Pre Specified Outcome: GammaH2AX Levels
Description: Wilcoxon test will be used to compare the percentage increase of gammaH2AX positive cells between the two treatment groups.
Time Frame: Up to 5 years
Reporting Status: Not Posted

8. Other Pre Specified Outcome: MGMT Expression, Assessed by Immunohistochemistry
Description: Results will be expressed as binary variables. Associations with objective response, with progression free survival and with overall survival will be tested using Fisher's exact test and log-rank test, respectively.
Time Frame: Up to 5 years
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Number of Circulating Tumor Cells
Description: The number of CTCs will be correlated with PFS and OS using Cox proportional hazards model. The change in CTCs will be correlated with radiographic response. The number of CTCs at baseline will be correlated with patient characteristics (disease burden, location of metastases, and progression at existing sites or new sites of disease). The number of CTC will be explored as a continuous variable and the presence of a threshold predictive of the outcome will be investigated.
Time Frame: Up to 5 years
Reporting Status: Not Posted

10. Other Pre Specified Outcome: PARP-1 Expression
Description: as for outcome 5
Time Frame: Up to 5 years
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Presence of MGMT Promoter Methylation, Assessed by the EpiTyper Assay
Description: as for outcome 8
Time Frame: Up to 5 years
Reporting Status: Not Posted

12. Other Pre Specified Outcome: PTEN Expression, Assessed by Immunohistochemistry
Description: as for outcome 5
Time Frame: Up to 5 years
Reporting Status: Not Posted

13. Other Pre Specified Outcome: RAD51 Expression, Assessed by Immunohistochemistry
Description: as for outcome 5
Time Frame: Up to 5 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Arm I (Veliparib and Temozolomide) | Arm II (Placebo and Temozolomide)
All-Cause Mortality (participants affected / at risk) | 41/52 | 39/45
Serious Adverse Events (participants affected / at risk) | 22/52 | 18/45
Other Adverse Events (participants affected / at risk) | 6/52 | 35/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Veliparib and Temozolomide) (N=52) | Arm II (Placebo and Temozolomide) (N=45)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Anorexia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dehydration (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Fatigue (General disorders) | 0 (0) | 1 (1)
Gastric perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Heart failure (Cardiac disorders) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Neoplasms ben/mal/unk (inc cyst/polyp) Other, spec (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (3)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2)
Anemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Appendicitis perforated (Gastrointestinal disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fall (Ear and labyrinth disorders) | 1 (2) | 0 (0)
Febrile Neutropenia (Investigations) | 3 (3) | 0 (0)
Gait disturbance (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Hepatic failure (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hip fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lung infection (Respiratory, thoracic and mediastinal disorders) | 2 (5) | 0 (0)
Nervous system disorders - Other, specify (Nervous system disorders) | 3 (3) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 5 (5) | 0 (0)
Sepsis (General disorders) | 2 (2) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
White blood cell decreased (Investigations) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Veliparib and Temozolomide) (N=52) | Arm II (Placebo and Temozolomide) (N=45)
Febrile neutropenia (General disorders) | 3 | 0
Nervous system disorders - Other, specify (Nervous system disorders) | 3 | 0
Platelet count decreased (Blood and lymphatic system disorders) | 5 | 14
Alanine aminotransferase increased (Blood and lymphatic system disorders) | 0 | 8
Alkaline phosphatase increased (Metabolism and nutrition disorders) | 0 | 6
Anemia (Blood and lymphatic system disorders) | 0 | 18
Anorexia (General disorders) | 0 | 3
Aspartate aminotransferase increased (Blood and lymphatic system disorders) | 0 | 3
Fatigue (General disorders) | 0 | 13
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 14
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 5
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 7
Lymphocyte count decreased (Blood and lymphatic system disorders) | 0 | 23
Nausea (General disorders) | 0 | 3
Neutrophil count decreased (Blood and lymphatic system disorders) | 0 | 6
White blood cell decreased (Blood and lymphatic system disorders) | 0 | 9
Creatinine increased (Metabolism and nutrition disorders) | 0 | 3
Hyponatremia (Metabolism and nutrition disorders) | 0 | 3
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 4
Lipase increased (Metabolism and nutrition disorders) | 0 | 4
Serum amylase increased (Metabolism and nutrition disorders) | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less